CLINICAL TRIAL: NCT03063541
Title: Prospective Randomized Open-label Trial to Evaluate Risk faCTor Management in Patients With Unruptured Intracranial Aneurysms
Brief Title: Acetylsalicylic Acid Plus Intensive Blood Pressure Treatment in Patients With Unruptured Intracranial Aneurysms
Acronym: PROTECT-U
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitätsmedizin Mannheim (Other)
Collaborators: UMC Utrecht (Other); Schwiete Stiftung, Mannheim, Germany (Unknown); KKS Netzwerk (Network); University of Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Nima Etminan, Vice Chair, Universitätsmedizin Mannheim
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PROTECT-U_V2.2_20_Feb_2017; 2017-000514-35 (EudraCT Number)
Record Dates: First submitted 2017-02-20; First posted 2017-02-24 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Unruptured Intracranial Aneurysms
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: controlled open trial, randomized 1:1
Who Masked: Outcomes Assessor
Masking Description: observer blinding
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acetylsalicylic acid, BP-target 120 (Experimental): 100 mg ASA plus intensified blood pressure management. Recommended systolic blood pressure 120 mm/Hg
  Interventions: Drug: Acetylsalicylic acid; Other: intensive blood pressure control
- standard care (No Intervention): blood pressure management according to guidelines

INTERVENTIONS:
Drug: Acetylsalicylic acid — 100 mg daily as one tablet
  Other Names: aspirin
  Arms: Acetylsalicylic acid, BP-target 120
Other: intensive blood pressure control — Patients are encouraged to seek any therapy to have a systolic blood pressure of 120 or below. They will be provided with a blood pressure measurement device and are advised to control blood pressure daily.
  Arms: Acetylsalicylic acid, BP-target 120

SUMMARY:
Purpose of this study is to assess the hypothesis that a strategy with acetylsalicylic acid (ASA) 100 mg/day, intensive blood pressure treatment (targeted systolic blood pressure below 120 mmHg), and a blood pressure measuring device reduces the risk of aneurysm rupture or growth compared with standard care (i.e. no ASA, blood pressure management according to standard blood pressure management, no blood pressure measuring device)

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older with an intradural, saccular unruptured aneurysm (UIA) in whom it is decided not to intervene with preventive endovascular or neurosurgical repair of the aneurysm and who are monitored on a regular base for aneurysm growth
* Last aneurysm imaging with either CTA/MRA/DSA within the last 3 months

Exclusion Criteria:

* All non-saccular UIAs or aneurysms related to arteriovenous malformations
* Frequent ASA use and/or indication for a vitamin K antagonist, or direct oral anticoagulant (DOAC) treatment at baseline
* Contra-indication for ASA
* History of hypersensitivity to ASA or to any other drug with similar chemical structure or to any excipient present in the pharmaceutical form of ASA
* Chronic kidney disease stage IV and V (GFR < 30 mL/min/1.73 m2)
* Pregnancy and lactation
* Participation in another clinical trial or observation period of competing trials, respectively
* Life-expectancy <3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 776 (Estimated)
Dates: Start 2017-09-21 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
aneurysm rupture or growth | 36 months
  aneurysm rupture (i.e. aneurysmal subarachnoid hemorrhage, SAH) or growth (increase in any aneurysm diameter by ≥1mm) on serial imaging (either two MR or CT angiographies)

SECONDARY OUTCOMES:
aneurysm volume | 36 months
  difference of aneurysm volume (in computerized measurements defined as increase of aneurysm volume in computerized measurements by >10% and >3mm3 or aneurysm shape (e.g. development of daughter sac)
new aneurysm | 36 months
  development of de novo aneurysm on serial imaging
therapy of aneurysm | 36 months
  clipping/coiling during the study period
stroke | 36 months
  any ischemic or haemorrhagic stroke, defined as clinical symptoms for stroke AND a compatible lesion on imaging
myocard infarction | 36 months
  myocardial infarction defined as increase of troponin, creatine-kinase MB and/or presence of new significant Q waves obtained in electrocardiography
vascular death | 36 months
  vascular death (including fatal stroke, fatal myocardial infarction, sudden death)
major bleeding | 36 months
  major spontaneous bleeding requiring hospitalisation defined as substantially disabling bleeding, intraocular bleeding leading to the loss of vision, or bleeding necessitating the transfusion of at least 2 units of erythrocyte concentrates
death | 36 months
  death from all other causes
achieved blood pressure | 36 months
  any data on blood pressure management used
Incidence of Treatment-Emergent Adverse and Serious Adverse Events | 36 months
  all adverse and serious adverse events related to the experimental intervention

CONTACTS AND LOCATIONS:
Overall Officials: Nima Etminan, PD Dr., Principal Investigator — UMM, Department of Neurosurgery; Mervyn D Vergouwen, MD,PhD, Principal Investigator — UMC Utrecht, Department of Neurology and Neurosurgery
Locations (18):
- Germany (12):
  - Department of Neurology and Neurosurgery, Goethe University, Frankfurt am Main, Hesse
  - Klinik für Neurochirurgie, Aachen
  - Neurochirurgische Klinik, Berlin
  - Neurochirurgische Klinik, Düsseldorf
  - Neurolgische Klinik, Erlangen
  - Klinik für Neurochirurgie, Essen
  - Klinik für Neurochirurgie, Göttingen
  - Klinik für Neurochirurgie, Hamburg
  - Neurologische Universitätsklinik, Heidelberg
  - Department of Neurosurgery, University Hospital Mannheim, Mannheim
  - Neurochirurgische Klinik und Poliklinik, München
  - Universitätsklinikum Münster, Münster
- Netherlands (6):
  - AMC Department of Neurology, Amsterdam
  - UMCG, Groningen
  - Leiden University Medical Center, Leiden
  - Neurochirurgisch Centrum CWZ, Nijmegen
  - Erasmus MC, Rotterdam
  - UMC, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vergouwen MD, Rinkel GJ, Algra A, Fiehler J, Steinmetz H, Vajkoczy P, Rutten FH, Luntz S, Hanggi D, Etminan N. Prospective Randomized Open-label Trial to evaluate risk faCTor management in patients with Unruptured intracranial aneurysms: Study protocol. Int J Stroke. 2018 Dec;13(9):992-998. doi: 10.1177/1747493018790033. Epub 2018 Jul 18. PMID 30019634